CLINICAL TRIAL: NCT05509257
Title: Development of a Pharmacodynamic Biomarker of Opioid Antagonism in Adolescents With Eating Disorders
Brief Title: Naltrexone Neuroimaging in Teens With Eating Disorders
Acronym: NN-RCT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephani Stancil, Assistant Professor, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00002228; K23MH130728 (NIH)
Record Dates: First submitted 2022-08-17; First posted 2022-08-22 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Eating Disorders; Binge Eating; Purging (Eating Disorders); Bulimia Nervosa; Anorexia Nervosa, Atypical
Keywords: Pediatric; Adolescent; Eating Disorder; Neuroimaging; Naltrexone; Pharmacodynamic Biomarker
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia; Bulimia Nervosa; Anorexia Nervosa | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): All participants will receive both naltrexone and placebo, separated by a washout period, in a randomized, crossover fashion. Those randomized to group A will receive naltrexone then placebo. Those randomized to group B will receive placebo then naltrexone.
  Interventions: Drug: Naltrexone; Drug: Placebo
- Group B (Experimental): All participants will receive both naltrexone and placebo, separated by a washout period, in a randomized, crossover fashion. Those randomized to group A will receive naltrexone then placebo. Those randomized to group B will receive placebo then naltrexone.
  Interventions: Drug: Naltrexone; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — Participants will receive a single oral dose in randomized, crossover fashion with a 2 week wash out period between interventions. Medication will be taken 2 hours prior the neuroimaging.
Drug: Placebo — Participants will receive a single oral dose of medication in randomized, crossover fashion with a 2 week wash out period between interventions.. Medication will be taken 2 hours prior the neuroimaging.

SUMMARY:
Using a randomized, placebo-controlled, crossover study, this study will evaluate functional magnetic resonance imaging (fMRI) as a pharmacodynamic biomarker of opioid antagonism in adolescents with eating disorders. The hypothesis is that fMRI will be able to detect acute reward pathway modulation by naltrexone (an opioid antagonist) in pre-defined regions of interest (anterior cingulate cortex, nucleus accumbens, dorsolateral prefrontal cortex).

DETAILED DESCRIPTION:
The investigators will use a randomized, placebo-controlled, double-blind, crossover trial to evaluate the use of fMRI as a pharmacodynamic biomarker of reward system modulation. The overall goal of this work is to develop an objective tool to detect acute drug response. If validated in future, larger trials, the pharmacodynamic biomarker may facilitate early phase/quantitative pharmacology studies of novel or repurposed agents expected to modulate the reward system. The reward system will be antagonized by naltrexone in adolescents aged 13-21 years with an ED defined by binge/purge behaviors (e.g., Anorexia Nervosa-Binge Purge, Bulimia Nervosa, Binge Eating Disorder). A crossover design was chosen to quantify within-individual change in opioid reward pathway modulation following antagonism. Eligible patients will be randomly assigned to Group A or Group B. A statistician (or other non-study staff) will generate the schedule and communicate with the investigation drug service to maintain the double-blind design. A washout period of at least 14 days will exceed the 48-hour carry-over effect from naltrexone 50 mg administered orally. The two study visits will be mirrored in structure and duration to maintain blinding.

It is not the intent of this study to generate data for submission to the FDA or to support a significant change in advertising of the drug. Storage, control and dispensation of the drug will occur through collaboration with the investigational drug service (IDS) pharmacy. Use of naltrexone for this study meets criteria for investigational new drug (IND) exemption, category #1 (21 Code of Federal Regulations (CFR) 312.2(b)(1)).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults aged 13-21 years
* Eating disorder diagnosis characterized by binge eating and/or purging (eg, Anorexia Nervosa-Binge/Purge, Bulimia Nervosa, Binge Eating Disorder, Other Specified Feeding/Eating Disorder) using Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria.
* Stable medication regimen (no dose or drug changes in the past 4 weeks)
* Participant and parent/legal guardian (if under 18 years) are willing and able to provide informed permission/assent/consent for the study

Exclusion Criteria:

* Pregnant (via UCG)
* Prior hypersensitivity reaction to naltrexone (e.g., anaphylaxis)
* Non-removable metal in the body that is magnetic resonance imaging incompatible
* Current naltrexone use
* Self-reported opioid use in the past 7 days
* A language barrier (e.g., non-English speaking) for the participant that precludes communication and/or ability to complete all study-related requirements.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Response | 2 hours post medication (naltrexone or placebo)
  Acute %Blood oxygenation level dependent (BOLD) change placebo vs. naltrexone in pre-defined regions of interest (anterior cingulate cortex, nucleus accumbens, dorsolateral prefrontal cortex)

SECONDARY OUTCOMES:
Maximum Concentration in Plasma (Cmax) | Blood sampled 0-7 hours post medication
  Naltrexone systemic exposure defined by the pharmacokinetic parameter Cmax
Area Under the Plasma Concentration vs. Time Curve (AUC) | Blood sampled 0-7 hours post medication
  Naltrexone systemic exposure defined by the pharmacokinetic parameter AUC

CONTACTS AND LOCATIONS:
Overall Officials: Stephani Stancil, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Research Institute, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stancil SL, Brewe ME, Tumberger J, Bartkoski M, Burns A, Yeh HW, Brucks MG, Bartolotti J, Voss M, Strawn JR, Abdel-Rahman S, Davis A, Brooks WM, Martin LE. Development of a pharmacodynamic biomarker of opioid antagonism in adolescents with eating disorders: Study protocol for the naltrexone neuroimaging randomized controlled trial (NN-RCT). Contemp Clin Trials. 2025 May;152:107874. doi: 10.1016/j.cct.2025.107874. Epub 2025 Mar 3. PMID 40043750